CLINICAL TRIAL: NCT03359889
Title: Post Marketing Surveillance Program of Praxbind Use in India.
Brief Title: PraxbindTM India PMS Program
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1321-0023
Record Dates: First submitted 2017-11-28; First posted 2017-12-02 (Actual); Results first posted 2021-02-16 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Thromboembolism
MeSH Terms: conditions — Thromboembolism | interventions — idarucizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients administered with PraxbindTM
  Interventions: Drug: PraxbindTM

INTERVENTIONS:
Drug: PraxbindTM — Drug
  Other Names: PRAXBIND, Praxbind, Prizbind

SUMMARY:
This program will be initiated after the commercial availability of PraxbindTM in India. It will include patients administered with PraxbindTM into the surveillance program after commercial availability in 2 years at selected centres approved by the regulatory authority.

ELIGIBILITY:
Inclusion Criteria:

- Patients treated with Pradaxa (dabigatran etexilate) capsules with requirement of rapid reversal of the anticoagulant effects of dabigatran: For emergency surgery/urgent procedures (or) In life-threatening or uncontrolled bleeding

- Written informed consent in accordance with International Conference on Harmonization Good Clinical Practice (GCP) guidelines and local legislation and/or regulations

Exclusion Criteria:

-Participation in a PraxbindTM clinical trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients, who receive PraxbindTM prescribed as per the approved label
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2018-12-26 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2020-01-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- India (3):
  - Mazumdar Shaw Medical centre, Bangalore
  - Columbia Asia Referral Hospital, Bengaluru
  - Care Hospital, Hyderabad

IPD SHARING:
Plan to Share IPD: Undecided
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions: 1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). Requestors can use the following link http://trials.boehringer-ingelheim.com/ to:
  1. find information in order to request access to clinical study data, for listed studies.
  2. request access to clinical study documents that meet criteria, and upon a signed 'Document Sharing Agreement.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter, non-interventional, drug administration surveillance program.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Praxbind®: Patients in a clinical practice setting treated with Pradaxa® (dabigatran etexilate) capsules with requirement of rapid reversal of the anticoagulant effects of dabigatran were treated with idarucizumab (Praxbind®). 1 vial of 50 milliliter (ml) contains 2.5 gram (g) idarucizumab (50 milligram/milliliter) given as an intravenous (IV) infusion, total recommended dose of 5 g.
Period: Overall Study
Arm/Group | Praxbind®
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Treated Set: Includes patients, who signed the ICF (Informed consent form), met the eligibility criteria and received Praxbind®.
Arm/Group | Praxbind®
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (8.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Suspected Adverse Drug Reactions (ADRs) and Fatal Adverse Events (AEs)
Description: Number of participants with suspected adverse drug reactions (ADRs) and fatal adverse events (AEs) occurring within 7 days after Praxbind® administration.
Time Frame: Up to 7 days following treatment.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Praxbind®
Number analyzed (Participants) | 5
Participants
  Number of participants with ADRs | 0
  Number of participants with AEs | 0

2. Secondary Outcome: Percentage of Patients Who Received Praxbind® Either for Emergency Surgery/Urgent Procedures or for Life-threatening or Uncontrolled Bleeding
Description: Percentage of patients who received Praxbind® either for emergency surgery/urgent procedures or for life-threatening or uncontrolled bleeding.
Time Frame: Data collected from patients who had been treated with Praxbind® within 2 years of the commercial availability of Praxbind®.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Praxbind®
Number analyzed (Participants) | 5
Percentage of participants
  For emergency surgery/urgent procedures | 20
  In life-threatening or uncontrolled bleeding | 80

ADVERSE EVENTS:
Time Frame: Up to 7 days following treatment.
Description: Treated Set: Includes patients, who signed the ICF (Informed consent form), met the eligibility criteria and received Praxbind®.
Arm/Group | Praxbind®
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 1/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Praxbind® (N=5)
Abdominal pain (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-03-23): https://cdn.clinicaltrials.gov/large-docs/89/NCT03359889/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-11): https://cdn.clinicaltrials.gov/large-docs/89/NCT03359889/SAP_001.pdf